CLINICAL TRIAL: NCT04901481
Title: Pilot Evaluation of the Empower Neuromodulation System for Anxiety Treatment
Brief Title: Empower Neuromodulation System - Pilot Study for Anxiety Treatment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to fully enroll study.
Sponsor: Theranova, L.L.C. (Industry)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRD-12-1396-01; R43AT011497 (NIH)
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-04

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Intervention Model Description: At enrollment, participants will be randomized (1:1) to receive either the active or sham treatment for the duration of the 6-week study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Research staff will not provide any details that would cause participants to become unblinded to the treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active treatment (Experimental): Participants will self-administer treatment with the Empower device at the active treatment anatomic location twice daily for six weeks. Treatment adherence will be assessed and participants will complete surveys to evaluate the feasibility and acceptability Empower active treatment.
  Interventions: Device: Empower Neuromodulation System
- Sham treatment (Sham Comparator): Participants will self-administer treatment with the Empower device at the sham treatment anatomic location twice daily for six weeks. Treatment adherence will be assessed and participants will complete surveys to evaluate the feasibility and acceptability Empower sham treatment.
  Interventions: Device: Empower Neuromodulation System

INTERVENTIONS:
Device: Empower Neuromodulation System — Peripheral nerve stimulation with the Empower device. The active and sham treatments only differ by the location of application on the body.

SUMMARY:
This study evaluates the effects of peripheral nerve stimulation on anxiety levels in participants with Generalized Anxiety Disorder (GAD). This is a pilot investigation in which participants will randomized (1:1) to the active or sham treatment.

DETAILED DESCRIPTION:
Generalized anxiety disorder (GAD) is a chronic, recurring condition that affects approximately 6.4 million American adults each year. GAD is one of the most common anxiety disorders and is costly to treat. First-line treatments for GAD include medication (e.g. SSRIs, SNRIs), cognitive behavioral therapy, or both in combination. Peripheral nerve stimulation via acupuncture has been shown to directly decrease clinical anxiety scores. The investigators have developed the Empower Neuromodulation System, a non-invasive, portable transcutaneous electrical nerve stimulation (TENS) device intended to stimulate peripheral nerves for the treatment of anxiety. In this study, a randomized, controlled study will be conducted in participants with GAD. Participants will self-administer twice daily treatments with the Empower device. In this pilot study, the primary endpoints will be feasibility and acceptability, with safety and effectiveness evaluated as exploratory endpoints.

ELIGIBILITY:
Inclusion Criteria:

* ≥19 years old
* Current diagnosis of GAD per DSM-5 via M.I.N.I. assessment by clinician
* Hamilton Anxiety Rating Scale (HAM-A) ≥18
* Negative urine pregnancy test at screening (females only)
* Able to provide informed consent
* Capable and willing to follow all study-related procedures

Exclusion Criteria:

* Has current (past 30 days) psychotic or bipolar disorder, homicidal ideation, psychiatric hospitalization, or moderate/severe substance use disorders per clinician assessment via M.I.N.I.
* Hamilton Depression Rating Scale (HAM-D) ≥18
* PTSD Checklist for DSM-5 (PCL-5) ≥51
* Exhibits suicidal intent as confirmed on the Columbia-Suicide Severity Rating Scale-Revised (C-SSRS-R) with a "Yes" response to question 4 or question 5 or to question 6 in the past 3 months.
* Changes in psychoactive medications in the past 30 days (including but not limited to psychotropic medications, thyroid hormone medication, steroids), with the exception of benzodiazepines
* If regularly taking benzodiazepines, has had changes in benzodiazepine dosing in the past 30 days or average use >2 days per week
* Psychotherapy was initiated or discontinued in the past 30 days or psychotherapy modality was changes in the past 30 days
* Has a history of epilepsy or a seizure disorder
* Has been diagnosed with peripheral nerve damage of the arm or hand or has numbness or tingling in the arm or hand at least weekly
* Is currently pregnant or breastfeeding, has been pregnant within the past 6 months or intends to become pregnant during the study period
* Currently has an active implant and/or an electrical or neurostimulator device, including but not limited to cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, sacral stimulator, bone growth stimulator, or cochlear implant
* Has an electrically conductive metal object (e.g. jewelry) that cannot be removed from the upper extremities and will directly contact the gel electrodes of the Empower Neuromodulation System at the active or sham anatomic location
* Has an open incision, wound, scar, active infection or otherwise compromised skin that will directly contact the gel electrodes of the Empower Neuromodulation System at either the active or sham anatomic location
* Does not have daily access to an electrical outlet for charging the investigational device and associated smartphone
* Has used of an investigational drug/device therapy within the past four weeks
* Unable to provide informed written consent
* Has any medical condition that would, in the opinion of the investigator, make the participant ineligible

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Burnett, MD, Principal Investigator — TheraNova, LLC
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bang, Heejung et al. "Blinding assessment in clinical trials: A review of statistical methods and a proposal of blinding assessment protocol." Clinical Research and Regulatory Affairs 27 (2010): 42 - 51.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 participants signed the Informed Consent Form and screened. 12 Subjects were fully enrolled.
Pre-assignment Details: Of 18 subjects that signed the Informed Consent, 6 did not meet all of the Inclusion/Exclusion criteria before randomization to a study arm. Therefore, only 12 subjects were fully enrolled and randomized into the trial.
Period: Overall Study
Arm/Group | Active Treatment | Sham Treatment
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Sham Treatment | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 44 [25 to 56] | 41 [26 to 59] | 41 [25 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 3 | 6 | 9
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Treatment Adherence
Description: Feasibility as assessed via treatment adherence (treatment sessions administered as a percentage of total possible) for each participant
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage of Treatment Sessions
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 6 | 6
Percentage of Treatment Sessions | 82 (19) | 72 (29)

2. Primary Outcome: Usability
Description: Acceptability as assessed via a usability assessment (System Usability Scale (SUS)). For the SUS, the score range is 0 to 100, with a higher score indicating the stimulation system's better usability. The survey includes 10 questions in which statements about the system are rated from "Strongly disagree" up to "Strongly agree".
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 6 | 6
Units on a scale | 73 (19) | 77 (19)

3. Secondary Outcome: Effective Nerve Stimulation
Description: The percentage of treatment sessions that provide effective nerve stimulation as assessed via participant-reported confirmation of tingling sensation
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: % of treatments that felt skin tingling
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 6 | 6
% of treatments that felt skin tingling | 98 (2) | 100 (1)

4. Secondary Outcome: Satisfaction With Treatment
Description: The overall satisfaction with treatment (via 100-mm Visual-Analog Scale (VAS)). For the VAS, the score range is 0 to 100, with a higher scoring meaning higher satisfaction.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: VAS score
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 6 | 6
VAS score | 52 (25) | 42 (22)

5. Secondary Outcome: Number of Participants With Device-related Adverse Events
Description: Safety assessment via device-related adverse events
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 6 | 6
Participants | 0 | 1

6. Secondary Outcome: Change in Hamilton Anxiety Rating Scale (HAM-A) Score From Baseline to 6weeks
Description: Anxiety severity evaluation via clinician-administered Hamilton Anxiety Rating Scale (HAM-A) score. For the HAM-A, the score range is 0 to 56, with a higher scoring meaning more severe anxiety.
Time Frame: 6 weeks
Population: Change in HAM-A score from Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 6 | 6
Score | -6.0 (9.4) | -12.2 (4.5)

7. Secondary Outcome: Change in Participant-reported Beck Anxiety Inventory (BAI) Score From Baseline to 6 Weeks
Description: Anxiety severity evaluation via participant-reported Beck Anxiety Inventory (BAI) score from Baseline to 6 weeks. For the BAI, the score range is 0 to 63, with a higher scoring meaning more severe anxiety.
Time Frame: 6 weeks
Population: Change in BAI score from Baseline to 6 week visit
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 6 | 6
Score | -2.8 (9.4) | -2 (5.8)

8. Other Pre Specified Outcome: Participant Blinding to Treatment Group at 6 Weeks
Description: Participant blinding to treatment group will be assessed. All participants will be asked if they believe that they have received the real treatment, with possible responses of Yes, No, or Don't Know. Then, for the active and sham treatment groups, the blinding index will be calculated, where the blinding index can range from -1 to 1. A score of 1 means that all participants have guessed correctly about group assignment, a score of -1 means that all participants have guessed incorrectly about group assignment.
Time Frame: 6 weeks
Population: Blinding Index at 6 week visit
Measure: Mean (95% Confidence Interval); unit: Index
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 6 | 6
Index | -0.4 [-0.58 to -.22] | -0.17 [-0.40 to 0.07]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the nominal 6 weeks after enrollment.
Arm/Group | Active Treatment | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 1/6 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=6) | Sham Treatment (N=6)
Diarrhea (Infections and infestations) | 0 (0) | 1 (1) — Norovirus
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=6) | Sham Treatment (N=6)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0)
Nausia (Infections and infestations) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Burning sensation at site of electrodes (Product Issues) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT04901481/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT04901481/ICF_001.pdf